An Open-Label, Long-Term Safety and Tolerability Study of Depot Buprenorphine (RBP-6000) in Treatment-Seeking Subjects With **Study Title** 

Opioid Use Disorder

**NCT Number** NCT02510014

April 10, 2017 Date



# **Statistical Analysis Plan**

| Sponsor: | Indivior Inc. |
|---|---|
| Protocol No: | RB-US-13-0003 |
| Version No./Date | Amendment 4/04-Aug-2016 |
| Title | An Open-Label, Long-Term Safety and Tolerability Study of Depot Buprenorphine (RBP-6000) in Treatment-Seeking Subjects With Opioid Use Disorder |
| CRF Version<br>No./Date | 3.0 / 22-Sep-2016 |
| PRA Project Id: | RBU13003-130003 |
| SAP Version<br>No./Date: | 3.0 / 10-Apr-2017 |

## **Approvals**

| Chanas | |
|--------------------------|-----------------------------------------|
| Sponsor | |
| Sponsor Name: | Indivior Inc. |
| Biostatistics/ Title: | / Head of Data and Statistical Sciences |
| Signature /Date: | |
| Medical/Title: | / Clinical Research Physician |
| Signature /Date: | |
| Medical/Title: | / Medicines Development Lead |
| Signature /Date: | |
| PRA | |
| Project Manager/Title: | Project Director |
| Signature /Date: | |
| Biostatistician / Title: | / Biostatistician |
| Signature /Date: | |

PRS 005 T 17 E 



## **Table of Contents**

| Approvals | |
|-------------------------------------------------------------|----|
| Table of Contents | 2 |
| 1.0 Introduction | 4 |
| 1.1 Changes from Protocol | 4 |
| 2.0 Study Objectives | 4 |
| 2.1 Primary Objective | 4 |
| 2.2 Secondary Objectives | 4 |
| 2.3 Tertiary Objectives | 4 |
| 3.0 Study Design | 5 |
| 3.1 Sample Size Considerations | 6 |
| 3.2 Randomization | 6 |
| 3.3 Study Duration | |
| 4.0 Study Variables and Covariates | 7 |
| 4.1 Primary Variables | 7 |
| 4.2 Secondary Variables | 7 |
| 4.3 Tertiary Variables | 7 |
| 5.0 Definitions | 8 |
| 6.0 Analysis Sets | 11 |
| 6.1 All Screened Subjects | |
| 6.2 Run-In Safety Analysis Set | 12 |
| 6.3 Safety Analysis Set | 12 |
| 6.4 PK Analysis Set | |
| 7.0 Interim Analyses (Data Cut Review) | 12 |
| 8.0 Data Review | |
| 8.1 Data Handling and Transfer | 12 |
| 8.2 Data Screening | 12 |
| 9.0 Statistical Methods | 12 |
| 9.1 Subject Disposition | 13 |
| 9.2 Protocol Deviations | 13 |
| 9.3 Demographic and Baseline Characteristics | 13 |
| 9.3.1 Medical History | 14 |
| 9.3.2 Prior and Concomitant Medications | 14 |
| 9.4 Study Treatment Exposure | 14 |
| 9.5 Efficacy Analysis | 14 |
| 9.5.1 Self-reported and Urine Samples Illicit Drug Use | |
| 9.5.2 Clinical Opioid Withdrawal Scale (COWS) Total Score | 16 |
| 9.5.3 Subjective Opioid Withdrawal Scale (SOWS) Total Score | 16 |
| 9.5.4 Opioid Craving VAS Total Score | 16 |
| 9.6 Primary Safety Analyses | 17 |
| 9.6.1 Incidence of Adverse Events | 17 |
| 9.6.2 Laboratory Data | 19 |
| 9.6.3 Vital Signs | 20 |
| 9.6.4 Other Safety Variables | 20 |
| 9.7 Pharmacokinetic Analysis | 21 |
| 10.0 Validation | 21 |
| 11.0 References | 21 |





| Appendix 1 Glossary of Abbreviations | 22 |
|---|---|
| Appendix 2 List of Preferred Terms from Standard MedDRA Queries for Adverse Events | |
| Interest | |
| Appendix 3 List of Post-text Tables, Figures, Listings, and Supportive SAS Output Append | |



#### 1.0 Introduction

This statistical analysis plan (SAP) describes the statistical methods to be used during the final reporting and analyses of data collected for the full study (Protocol RB-US-13-0003).

This SAP should be read in conjunction with the study protocol and case report form (CRF). This version of the plan has been developed using the protocol dated 04AUG2016 and CRF dated 22SEP2016.

The SAP for study RB-US-13-0003 was developed in three stages. SAP Version 1.0was finalized so that programming could begin earlier in the process. SAP Version 2.0 was finalized before the interim database lock and was used for the interim anlaysis. This SAP version 3.0 will be finlaised and used for the final reporting and analysis of the full study data.

## 1.1 Changes from Protocol

The following changes to the analysis planned in the protocol were made:

- The addition of an analysis set (Run-In Safety Analysis Set) was made to aid in the analysis of the Run-In period.
- Electrocardiograms (ECGs) overall impression summaries will only be summarized by normal or abnormal; protocol says they should be summarized by normal, abnormal not clinically significant, or abnormal clinically significant, but there is no distinction of clinical significance for abnormal results.
- There will be no mixed-effect model for repeated measure analysis on the clinical outcome data, Clinical Opiate Withdrawal Scale (COWS), Subjective Opidate Withdrawal Scale (SOWS), and Opioid Craving Visual Analog Scale (VAS), due to the nature of the study design.
- The Clinical Outcome Assessment Analysis Set has been removed since this is a safety study.
- Total score for electronic Columbia Suicide Severity Rating Scale will not be summarized.
- Physical examination data is collected as a part of the corresponding safety assessment (i.e. adverse events (AEs), vital signs).

## 2.0 Study Objectives

Indivior Inc., formerly Reckitt Benckiser Pharmaceuticals Inc. (RBP) is developing RBP-6000, a long-acting formulation of buprenorphine for monthly subcutaneous (SC) injection, for the treatment of opioid use disorder (OUD).

## 2.1 Primary Objective

To assess the long-term safety and tolerability of RBP-6000 SC injections in subjects with opioid use disorder.

## 2.2 Secondary Objectives

To collect clinical outcome data with RBP-6000 SC injections in subjects with opioid use disorder.

## 2.3 Tertiary Objectives

To evaluate the:

- Pharmacokinetics (PK) of RBP-6000.
- Relationship between RBP-6000 PK and clinical outcome data, and
- Impact of RBP-6000 on health and economic outcomes.



A stand-alone SAP will be developed for the health and economic outcomes. PK will be reported separately from the clinical study report.

## 3.0 Study Design

This is a multicenter, open-label, long-term Phase III safety study in which approximately 600 subjects diagnosed with opioid use disorder will be enrolled (approximately 300 subjects who did not participate in the RB-US-13-0001 study [hereafter referred to as "de novo" subjects] and approximately 300 subjects that completed the RB-US-13-0001 study [hereafter referred to as "roll-over subjects")]. Subject participation will be based on the Investigator's determination that initiation or continuation of study treatment is appropriate; and, that among subjects who are continuing from the RB-US-13-0001 study, there have been no significant protocol deviations or clinically important AEs that would preclude inclusion of the subject in RB-US-13-0003.

Before receiving the first injection of RBP-6000 in this safety study, all subjects will undergo a Run-In period with SUBOXONE® (buprenorphine/naloxone) sublingual film to avoid precipitating a withdrawal syndrome and to preserve blind in subjects treated with placebo in the RB-US-13-0001 study. Subjects will be inducted onto SUBOXONE sublingual film consistent with the SUBOXONE sublingual film label; they will then complete a 1 to 11 day SUBOXONE sublingual film Dose Adjustment period.

Once subjects meet the criteria (on Day -11 to Day -1) of no significant opioid craving (≤20 mm on the Opioid Craving VAS and no significant withdrawal (≤12 on the COWS) they may receive the first SC injection of RBP-6000 (containing 300 mg of buprenorphine). Subjects with significant withdrawal signs/symptoms (defined as > 12 on the COWS) or significant cravings for opioids (defined as >20 mm on the Opioid Craving VAS) after the end of the 2-week SUBOXONE sublingual film Run-In period will not be eligible to continue in the study and will be referred for treatment.

On Day 1 of the study (initiation of study drug injections), all subjects will receive a SC injection of 300 mg of buprenorphine in RBP-6000. Subsequent doses of RBP-6000 may be adjusted down to 100 mg and back up to 300 mg based on the medical judgment of the Investigator. After injection of RBP-6000, subjects will not be permitted to receive supplemental SUBOXONE sublingual film during the RBP-6000 treatment period. Subjects who require supplemental SUBOXONE sublingual film or other sublingual buprenorphine pharmacotherapy during the RBP-6000 treatment period will be withdrawn from the study and referred for appropriate treatment.

Subjects will return to the clinic for monthly injection visits (every 28 -2/+4 days) for a total of up to 12 injections for *de novo* subjects or for a total of 6 injections for roll-over subjects. ECG recordings and vital signs will be collected pre and post each SC injection. All ECGs will be interpreted by a central monitoring facility. Subject-reported injection site pain VAS scores will be collected at various times up to 1 hour after each injection. Local injection site grading will be collected at various time points starting immediately after injection and will be evaluated for pain, tenderness, warmth, itching, erythema, inflammation or swelling, and bruising using a 4-point severity scale. At each visit after injections begin, the injection site will be assessed by site staff and will also be evaluated for evidence of attempts to remove the depot.

Subjects will need to return to the clinic weekly for the first 5 weeks and biweekly (i.e., every 2 weeks) until injection 6, and monthly for the rest of the study period for urine drug screens (UDS), Timeline Followback (TLFB) interviews, opioid craving VAS evaluation, COWS and subject reported outcomes (SOWS). Subjects will continue to receive counseling (manual-guided behavioral therapy) during the study. Safety assessments will be collected at each injection visit and/or at injection follow-up visits and will include the following: vital signs, electronic Columbia Suicide Severity Rating Scale (eC-SSRS) responses, ECGs, laboratory tests (hematology, chemistry, urinalysis, and pregnancy test), concomitant medications, and AEs.



Approximately 2 months prior to the scheduled end of study (EOS) visit, the subject's ongoing treatment options will be reviewed with the investigator. At the EOS, 2 transition treatment options may be offered if the subject is eligible:

- Subjects who complete RBP-6000 treatment period may be offered entry into an open label extension study of RBP-6000 (Study INDV-6000-301). Eligibility will be based on meeting the inclusion and exclusion criteria and the medical judgment of the Investigator.
- Subjects who do not meet the eligibility criteria of the extension study, or subjects who do not
  wish to enroll may alternatively enter a 4-week SUBOXONE transition period if deemed suitable
  by the investigator. Subjects should be dosed using the Investigators medical judgment. Any
  additional unscheduled visits required by the subject for the SUBOXONE transition will not be
  compensated by the Sponsor.

Subjects that did not enroll onto the INDV-6000-301 should be contacted by telephone approximately 4 weeks after EOS for a safety follow-up assessment of AEs and use of concomitant medications. The safety assessments used include evaluations of AEs, serious AEs (SAEs), discontinuations from study due to AEs; local injection site tolerability (e.g., injection site grading); injection site pain using a subject-reported VAS; suicidality using the eC-SSRS, concomitant medications; changes in clinical laboratory results; vital sign measurements; 12-lead ECGs, and physical examination results. The instruments used to measure clinical outcomes (e.g., COWS, SOWS, Opioid Craving VAS, and eC-SSRS) were developed to measure the specific symptoms exhibited by and the challenges facing opioid-dependent individuals.

## 3.1 Sample Size Considerations

This study is designed to assess the long-term safety, tolerability, and clinical outcomes of RBP-6000 SC injections in subjects with opioid use disorder. Approximately 300 *de novo* subjects as well as approximately 300 roll-over subjects who completed the RB-US-13-0001 study will be enrolled into this long-term safety study. The planned number of subjects was designed to ensure at least 100 subjects reach 1 year of treatment with RBP-6000 (as advised in the ICH-E1A Guideline – The Extent of Population Exposure to Assess Clinical Safety: For Drugs Intended for Long-term Treatment of Non-Life-Threatening Conditions).

#### 3.2 Randomization

This is an open-label study and does not involve randomization.

### 3.3 Study Duration

The expected maximum duration of participation for *de novo* subjects is up to approximately 55 weeks consisting of up to a 7-day screening period, up to a 14-day SUBOXONE sublingual film Run-In, up to a 48-week open-label treatment period, and a 4-week follow-up and transition period when subjects will receive the same dose of SUBOXONE that they received at Day -1 and their ongoing treatment options will be reviewed.

The expected maximum duration of participation for roll-over subjects is up to approximately 31 weeks, consisting of up to a 7-day screening period, up to a 14-day SUBOXONE sublingual film Run-In, a 24-week open-label treatment period, and a 4-week follow-up and transition period when they will receive the same dose of SUBOXONE that they received at Day -1 and their ongoing treatment options will be reviewed.

If at least 100 subjects reach 1 year of exposure to RBP-6000 in RB-US-13-0001 and RB-US-13-0003, the study may be stopped early, and all remaining subjects will complete EOS procedures and enter the SUBOXONE Transition Period/Safety Follow-up.

Subjects who receive at least 1 dose of RBP-6000 and discontinue the trial for any reason will be required to complete the Early Termination (ET) visit.

## 4.0 Study Variables and Covariates

## 4.1 Primary Variables

The following variables will be evaluated to assess the safety and tolerability of RBP-6000:

- Incidence of treatment-emergent adverse events (TEAEs).
- Changes in clinical laboratory results.
- Vital sign measurements.
- Other variables related to safety
  - 12-lead ECGs.
  - Medical history.
  - Suicidality using the eC-SSRS.
  - Prior and concomitant medications.
  - Local injection site tolerability (e.g., injection site grading).
  - Injection site pain using a subject-reported VAS.
  - Physical examination results.

## 4.2 Secondary Variables

The following secondary variables will be evaluated to analyze clinical outcomes:

- COWS total score.
- SOWS total score.
- Opioid Craving VAS total score.
- Self-reported illicit drug use.
- Percentage of negative urine drug screen samples.

## 4.3 Tertiary Variables

- PK of RBP-6000.
- Health economic and outcome data (to be analyzed in a separate SAP)
  - o Beck Depression Inventory.
  - Brief Pain Inventory.
  - EuroQoL EQ-5D-5L.
  - o 36-Item Short Form Health Survey.
  - Medication Satisfaction Questionnaire.
  - Healthcare Resource Utilization.
  - Treatment Effectiveness Assessment.
  - Addiction Severity Index Lite.

Statistical Analysis Plan

Effective Date: 10-Apr-2017 Version 3.0

Sponsor: Indivior Inc. Protocol no: RB-US-13-0003

#### 5.0 Definitions

#### Abstinent

A subject is defined as being abstinent from opdioid drug use if his/her UDS and TLFB results for opioids are negative.

#### Age

Age is defined as date of informed consent - date of birth + 1.

#### **Baseline and Change from Baseline**

Baseline is defined as the last non-missing value prior to SC injection of RBP-6000 on Day 1 of the RB-US-13-0003 study.

Change from baseline = (post-baseline value - baseline value).

#### **Completed Study**

A subject will be deemed to have completed the study if he/she has received 6 doses (roll-over) or 12 doses (de-novo) of RBP-6000 and completed the EOS visit.

#### **Clinical Opioid Withdrawal Scale Total Score**

The COWS total score is defined as the sum of the responses to the 11 questions including resting pulse rate, gastrointestinal upset, sweating, tremor, restlessness, yawning, pupil size, anxiety or irritability, bone or join aches, gooseflesh skin, and runny rose or tearing. Each answer to a corresponding question is assigned a value between 0 and 5. If 2 or more answers are missing, then a total score will be set to missing. If 1 question is missing, then the total score will be defined as the average of the non-missing responses multiplied by the total number of answered questions (hereafter referred to as normalized).

#### **Prior and Concomitant Medications**

Prior medications will be any medication taken before the date of first dose of SUBOXONE (during run-in) in the RB-US-13-0003 study.

Concomitant medications will be defined as any medication taken on or after the first dose of SUBOXONE (during run-in) in the RB-US-13-0003 study.

Concomitant medications include those medications that are ongoing at the time a subject rolls-over from the RB-US-13-0001 study. Medications or supplements that meet any of the following criteria will be considered concomitant:

- Missing both start and stop dates
- Having a start date prior to the start of first dose of SUBOXONE and missing the stop date
- Having a stop date after the first injection missing the start date.

#### **Subject Type**

Subjects will be categorized as either de novo or roll-over (from the RB-US-13-0001 study.

#### Treatment-emergent Adverse Events

TEAEs are those that started following the first dose of RBP-6000 in this study or were present prior to the first dose of RBP-6000 in this study regardless of causality and increased in severity following administration of RBP-6000 regardless of causality≤30 days after the last dose of RBP-6000. All AEs which change in severity or relationship to RBP-6000 are assigned a new start date and captured as a new AE. AEs include those events that are ongoing at the time a subject rolls-over from the RB-US-13-0001 but these events will not be considered treatment-emergent.



#### **Run-In Adverse Events**

An AE for the run-in period is an AE that either commenced during the run-in period or was present prior to the initiation of run-in, but increased in severity during run-in, regardless of causality, and prior to the first injection of RBP-6000.

#### **Outcome of Death**

Any AE with an outcome of fatal or study discontinuation due to death.

#### **Subjective Opioid Withdrawal Scale Total Score**

The SOWS total score is defined as the sum of the responses to the 16 questions as indicated by the subjects on how they feel at the time of completed the questionnaire including anxiousness, yawning, perspiring, teary eyed, runny nose, goosebumps, shaky, hot flushes, cold flushes, bones and muscle achiness, restlessness, nausea, vomiting, muscle twitching, stomach cramps, and feeling like using now. Each answer to a corresponding question is assigned a value between 0 and 4. If 3 or more responses are missing, then a total score will be set to missing. If less than 3 responses are missing, then the total score will be normalized.

#### Suicidal Ideation Scoring

The suicidal ideation score ranges from 0 to 5 and depends on the answers to the suicidal ideation portion of the eC-SSRS. The score is the maximum suicidal ideation category (in the following order: 1 = wish to be dead, 2 = Non-specific active suicidal thoughts, 3 = active suicidal ideation with any methods (not plan) without intent to act, 4 = active suicidal ideation with some intent to act, without specific plan, and 5 = active suicidal ideation with specific plan and intent) present at the assessment. If all answers to these questions are "No" then the suicidal ideation score is 0.

#### Suicidal Ideation Intensity Rating:

The suicidal ideation intensity rating is the sum of the five intensity item scores to create a total score (range 0 to 25). The five intensity items include frequency, duration, controllability, deterrents, and reason for ideation. Each item is scored from 0 to 5 with 5 representing the most severe intensity.

#### Suicidal Behavior Scoring

The suicidal ideation score ranges from 0 to 5 and depends on the answers to the suicidal behavior portion of the eC-SSRS. The score is the maximum suicidal ideation category (in the following order: 1 = preparatory acts or behavior, 2 = aborted attempt, 3 = interrupted attempt, 4 = actual attempt, and 5 if the subject has an AE with a preferred term of completed suicide. If all answers to these questions are "No" and the subject does not have an AE with a preferred term of completed suicide then the suicidal behavior score is 0.

#### **Treatment Duration (weeks)**

Treatment duration will be defined as (treatment stop date – treatment start date + 1)/7 where treatment stop date is defined as date of last RBP-6000 injection + 28 days.

Statistical Analysis Plan Effective Date: 10-Apr-2017 Version 3.0

Sponsor: Indivior Inc.
Protocol no: RB-US-13-0003

#### Percentage of Urine Drug Screen and Self-Report Results

Subjects' self-reported illicit drug use from the TLFB and results from the UDS will be combined into a single endpoint in the following manner:

- If both the TLFB and the UDS have a negative result at a particular visit, then the visit will be considered to have a negative result at that visit.
- If either the TLFB or UDS, or both, have a non-negative result at a particular visit, then the visit will be considered to have a non-negative result at that visit.

To be conservative, missing UDS or TLFB data will be imputed as non-negative.

| Urine Drug Screen Result for | Self-Report of Illicit Opioid Use | Overall |
|---|---|---|
| Opioids | Result | Result |
| Nonnegative | Nonnegative | Nonnegative |
| Nonnegative | Negative | Nonnegative |
| Negative | Nonnegative | Nonnegative |
| Negative | Negative | Negative |

#### Treatment Success

A subject is defined as a treatment success if ≥80% urine samples negative combined with self-reports negative.

#### Visit Window for Remapping of Early Termination visit

Duration will be derived in days as (ET visit date - treatment start date) + 1.

PRS 005 T 17 E 



#### Visit window for safety and efficacy assessments.

| Study Visit | Lower Window for Analysis<br>Day (ADY) | Upper Window for ADY |
|---|---|---|
| Week 1 Day 1 | 1 | 1 |
| Week 1 Day 2 | 2 | 5 |
| Week 2 Day 8 | 6 | 12 |
| Week 3 Day 15 | 13 | 19 |
| Week 4 Day 22 | 20 | 26 |
| Week 5 Day 29 | 27 | 38 |
| Week 7 Day 43 | 39 | 54 |
| Week 9 Day 57 | 55 | 68 |
| Week 11 Day 71 | 69 | 82 |
| Week 13 Day 85 | 83 | 94 |
| Week 15 Day 99 | 95 | 110 |
| Week 17 Day 113 | 111 | 122 |
| Week 19 Day 127 | 123 | 138 |
| Week 21 Day 141 | 139 | 166 |
| Week 25 Day 169 | 167 | 194 |
| Week 29 Day 197 | 195 | 222 |
| Week 33 Day 225 | 223 | 250 |
| Week 37 Day 253 | 251 | 278 |
| Week 41 Day 281 | 279 | 306 |
| Week 45 Day 309 | 307 | 335 |

If an ET visit/assessment happens any time between Day 1 and prior to End of Study visit, the following approach (Table) should be adopted to remap those ET visit to applicable study visit week based on the ADY variable value, defined as date of assessment – date of first dose + 1, of the ET date variable.

If Lower Window <= ADY (of ET date) <= Upper window, then set appropriate AVISIT value based on the above CRF study visits.

After re-mapping the ET visits to any of study visit weeks, if there are multiple records falling within the same week window, latest one with non-missing result will be flagged in analysis datasets and considered for analysis of by visit summary tables and figures.

## 6.0 Analysis Sets

## 6.1 All Screened Subjects

All screened subjects include any subject who signed the informed consent form.



Statistical Analysis Plan Effective Date: 10-Apr-2017 Version 3.0

Sponsor: Indivior Inc.
Protocol no: RB-US-13-0003

## 6.2 Run-In Safety Analysis Set

The Run-In Safety Analysis Set will include all subjects who received at least 1 dose of SUBOXONE during the Run-In period of the study.

## 6.3 Safety Analysis Set

The Safety Analysis Set comprises all subjects who received at least 1 dose of RBP-6000 during the openlabel treatment period of the study. This analysis set will be used for all safety analyses.

## 6.4 PK Analysis Set

The PK Analysis Set will include any subject who receives a dose of RBP-6000 or at least 1 dose of SUBOXONE sublingual film and has at least 1 PK sample collected post-dose.

## 7.0 Interim Analyses (Data Cut Review)

An interim safety analysis was conducted using all data up to and including the 12<sup>th</sup> August 2016. The data was anlysed and reported as per SAP version 2.0.

## 8.0 Data Review

## 8.1 Data Handling and Transfer

All of the data will come from the PRA Health Sciences data management group in SAS® dataset format (SAS version 9.4 or later) converted to Study Data Tabulation Model (SDTM) using SDTM Implementation Guide (SDTMIG) Version 3.1.3. Please refer to the Data Quality Plan for details.

The following vendors will be providing data for the study:

- WCT: PK data:
- ACM: Central laboratory data;
- ERT: SOWS, COWS, Opioid Craving VAS, Injection site grading scale, TLFB results, injection pain VAS, end time of the injections, and eC-SSRS data;
- Cardiocore: ECG data.

#### 8.2 Data Screening

Beyond the data screening built into the Data Management Plan, the programming of analysis datasets, tables, figures, and listings (TFLs) provides additional data screening. Presumed data issues will be output into SAS logs identified by the word "Problem" and extracted from the logs by a SAS macro and sent to PRA Data Management.

Review of a pre-data cut subset TFL run allows for further data screening prior to lock. The pre-data cut subset TFLs will be discussed with the sponsor in a data review meeting to identify any final data issues and seek corrections prior to database lock for the interim lock and final lock. The PRA statistician and the sponsor must approve final database lock.

#### 9.0 Statistical Methods

All statistical analyses will be performed using SAS® Version 9.4 or higher.

Categorical variables will be summarized using counts and percentages. Percentages will be rounded to one decimal place; except 100% will be displayed without any decimal places and percentages will not be displayed for zero counts. When assessments are not applicable (ie Post injection 6 visits for roll-over subjects), an N/A will displayed instead of a zero,



Continuous variables will be summarized using the number of observations (n), mean, standard deviation (SD), median, minimum, and maximum. The minimum, maximum, and 95% CI values (in some instances) will be displayed to the same level of precision as the raw data, the median and mean to one additional decimal place and the SD to two additional decimal places. The maximum number of decimal places will be 4. All summaries will be presented by subject type (de novo or roll-over) unless otherwise stated.

Unless otherwise stated, summaries will be presented by subject type (*de novo* or roll-over and total). Missing values will be presented by blank spaces. For partially missing dates, the information present will be printed; e.g., "--JAN2000".

For dichotomous outcome measures such as urine drug screen results (negative; non-negative) and self-reports for illicit opioid use (negative; non-negative), any missing observation will be set equal to "non-negative." Missing results for substances other than opioids will not be imputed. For all continuous endpoints (e.g., COWS, SOWS, and VAS), the missing data will not be imputed.

Only scheduled assessments per protocol Amendment 4 will be presented in tables and figures except for worst case post-baseline and at any time types of analyses (all post-baseline including unscheduled assessments data will be considered for this derivation) but all data will be presented in the listings.

#### 9.1 Subject Disposition

The number and percentage of all screened subjects in each analysis set will be summarized (de-novo, roll-over and total).

A summary of the number and percentage of all screen and enrolled subjects (de-novo, roll-over, total) at each center will be presented, including those centers who screened or enrolled no subjects.

The number and percentage of subjects screened, screen failures, entered the Run-In period, Run-In failures (including those who prematurely discontinued during the Run-In period), entered the RBP-6000 treatment period (i.e. received at least 1 dose of RBP-6000), and who completed the study will be presented, together with the number and percentage of subjects who prematurely discontinued from the RBP-6000 treatment period or in the Run-In period prematurely and a breakdown of the corresponding reasons for study discontinuation separately in each period.

A listing of all subjects' analysis set inclusions, disposition, and reasons for study discontinuation will be presented.

A listing of the inclusion/exclusion reasons for screen failure will be provided.

#### 9.2 Protocol Deviations

A listing of subjects in the Safety Analysis Set with important protocol deviations (PDV) will be provided. An important deviation is defined as:

- · Subject consent was never obtained
- Inclusion/Exclusion/Enrollment Criteria were violated

## 9.3 Demographic and Baseline Characteristics

Demographic and baseline characteristics (sex, ethnicity, race, age [years and categories of  $\geq$ 18-<30,  $\geq$ 30-<45,  $\geq$ 45-<60,  $\geq$ 60, and  $\geq$ 65], weight [kg], height[cm], waist-to-hip ratio, body mass index [BMI; kg/m²], tobacco use [never, former, current], caffeine use [never, former, current], alcohol use [never, former, current]) will be summarized by subject type (de novo, roll-over and total) using descriptive statistics for subjects in the Safety Analysis Set. Qualitative variables (sex, ethnicity, race, age categories, tobacco use, caffeine use, alcohol use) will be summarized using frequencies while quantitative variables (age, weight, height, BMI, waist-to-hip ratio) will be summarized using mean, SD, median, minimum, and maximum. Demographic and baseline data will also be listed for all screened subjects.



A further summary of the subjects will be presented for subgroups including opioid users at screening [injectable vs. non-injectable] and use of opioids during the Run-In period as indicated by a nonnegative UDS in the Safety Analysis Set.

History of drug use will be presented by substance and previous use for subjects in the Run-In Safety Analysis Set. All drug use history collected on the CRF will be listed including days of opioid drug use in the past 30 days, years of regular drug use in lifetime, and route the substance was administered for all screened subjects.

#### 9.3.1 Medical History

Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA) version 17.1 and summarized by the number and percentage of subjects in each system organ class (SOC), preferred term (PT), and subject type in the Safety Analysis Set.

Listings of medical history events for subjects in the Run-In Safety Analysis Set will be provided.

#### 9.3.2 Prior and Concomitant Medications

Medications received prior to exposure to SUBOXONE, categorized by preferred name and ATC level 4 class according to World Health Organization Drug Dictionary (WHODRUG; Version 2014SEP01DDE), will be summarized for the Safety Analysis Set. The number and percentage of subjects using each medication will be displayed together with the number and percentage of subjects using at least one medication. Additionally, medications received concomitantly with study will be summarized in the same manner for the Safety Analysis Set.

All prior and concomitant medications will be presented in separate listings for the Safety Analysis Set.

## 9.4 Study Treatment Exposure

A summary of the exposure to SUBOXONE during the Run-In period will be summarized by Run-In period (induction/dose adjustment), visit, administration/dispensation, and dosage for the Run-In Safety Analysis Set. A listing of SUBOXONE exposure (administration/dispensation) will be provided.

Exposure will be derived as date of first RBP-6000 injection on the RB-US-13-0003 study, to 28 days after the last RBP-6000 injection on this study.

The duration of exposure in the 0-<4 weeks through 48 - <52 weeks, total number of RBP-6000 doses received, the total number of actual doses as a continuous summary, and the total number of actual doses as a categorical summary will be presented for the Safety Analysis Set. RBP-6000 exposure data will also be listed detailing the dose of RBP-6000 received at each injection and the number of days between injections.

The number of subjects who have early removal of the RBP-6000 depot by physician will be presented for the Safety Analysis Set. Early removal of the study drug depot data including the reason and removal date and time will be listed.

## 9.5 Efficacy Analysis

All efficacy endpoints will be summarized for the Safety Analysis Set.



## 9.5.1 Self-reported and Urine Samples Illicit Drug Use

#### **Urine Drug Screen Result**

A subject will be deemed to have a 'non-negative' result for opioids when his/her urine drug screen result is greater than the upper limit of normal for any of the opioid drugs tested (Section 9.6.2.4).

#### Opioid Drug Classification (UDS)

| Drug | Opioid? |
|----------------------------|---------|
| Amphetamine | No |
| Barbiturates | No |
| Benzodiazepine | No |
| Benzoylecgonine | No |
| Buprenorphine <sup>1</sup> | No |
| Cannabinoids | No |
| Codeine | Yes |
| Hydrocodone | Yes |
| Hydromorphone | Yes |
| Methadone | Yes |
| Morphine | Yes |
| Opiate | Yes |
| Oxycodone | Yes |
| Oxymorphone | Yes |
| Phencyclidine | No |

<sup>&</sup>lt;sup>1</sup> Buprenorphine urine testing for de novo subjects was only included during the screening period; and urine testing for buprenorphine during the screening period was subsequently removed from the protocol per protocol amendment #1. The only subjects who tested positive during screening (when RBP-6000 was not being administered) were de novo subjects. Roll-over subjects were not tested for buprenorphine during screening. Neither de novo nor roll-over subjects were tested for buprenorphine at baseline or post-RBP-6000 administration.

#### Opioid Drug Classification (TLFB)

| Drug | Opioid? |
|------------------------------------|---------|
| Amphetamine/Methadone <sup>1</sup> | Yes |
| Barbiturates | No |
| Benzodiazepine | No |
| Buprenorphine | Yes |
| Cocaine | No |
| Ethanol | No |
| Methadone | Yes |
| Opioids | Yes |
| PCP | No |

<sup>&</sup>lt;sup>1</sup> The TLFB interview called for an assessment of the use of amphetamine/methamphetamine. However, the ePRO tablet was programmed to ask for the use of amphetamine/methadone. As a result, the primary analysis for the TLFB question of amphetamine/methadone will be assumed to be non-negative. A sensitivity analysis will be performed where the answer to the TLFB question of amphetamine/methadone of 'Use" will be assumed to be negative.

Subjects' self-reported illicit drug use from the TLFB and opioid detection from the UDS will be summarized together by showing the number and percentage of subjects who have  $\geq 0$ ,  $\geq 10\%$ ,  $\geq 20\%$ ,  $\geq 30\%$ ,  $\geq 40\%$ ,  $\geq 50\%$ ,  $\geq 60\%$ ,  $\geq 70\%$ ,  $\geq 80\%$ ,  $\geq 90\%$ ,  $\geq 100\%$  negative result and a continuous summary of the percent negative. The cumulative distribution function (CDF) of the percentage abstinence (negative self-reports from the TLFB combined with negative UDS for opioid use) will be presented in a graph. The graph will present the proportion of subjects who remained at least a given percentage abstinent from opioid drug



use, as defined in <u>Section 5</u>; for example, 10% on the x-axis represents the proportion of subjects who had at least 10% of their self-reported opioid drug use combined with UDS as abstinent.

Additionally, a table showing the percentage of subjects with negative results at each visit will be provided.

All missing results for opioids were considered nonnegative for opioids. Opioids non-negative indicates detection of buprenorphine (only self-reports), codeine, hydrocodone, hydromorphone, methadone, morphine, opiates, oxycodone, and oxymorphone in the urine drug screen and reporting of amphetamine/methadone, buprenorphine, methadone, and opioids use in the timeline followback.

The number and percentage of subjects abstinent between visits will be summarized by subject type for the Safety Analysis Set. Additionally, the time to first urine sample non-negative or TLFB self-report of non-negative for opioids will be analyzed in the Safety Analysis Set for subjects who are Abstinent on Day 1 using Kaplan-Meier analysis methods to determine the first quartile (25%) and median (days) along with their corresponding confidence intervals in each subject type and overall. Subjects who are abstinent throughout the trial will be censored on the date of their last negative urine sample of TLFB self-report for opioids.

The number and percentage of subjects who have a non-negative result in each substance tested in the UDS will be reported by subject type in the Safety Analysis Set. Additionally, the number and percentage of subjects at each visit who tested non-negative for non-opioid substances will be summarized by subject type in the Safety Analysis Set in a tables and in figures for amphetamine, barbiturates, benzodiazepine, cannabinoids, and phencyclidine.

Opioid TLFB and UDS results will be listed together. Additionally, all drugs identified in the TLFB interviews and detected in the UDS will be listed separately for the Safety Analysis Set.

## 9.5.2 Clinical Opioid Withdrawal Scale (COWS) Total Score

COWS total scores will be summarized by clinical visit and subject type using descriptive statistics (mean, median, SD, minimum, and maximum), including change from baseline. A listing of the COWS assessment will be provided for the Safety Analysis Set. Additionally, separate listings for the actual values (individual responses and total scores) and the change from baseline in total COWS score will be presented for the Safety Analysis Set.

A figure for the COWS scores over time will be created for all subjects in the Safety Analysis Set. An additional table and figure will be created for the Safety Analysis Set excluding subjects using illicit opioids (either by UDS or TLFB) at any time during the study.

#### 9.5.3 Subjective Opioid Withdrawal Scale (SOWS) Total Score

SOWS total scores will be summarized using descriptive statistics (mean, median, SD, minimum, and maximum), including change from baseline. A listing of the SOWS assessment will be provided for the Safety Analysis Set. Additionally, separate listings for the actual values (individual responses and total scores) and the change from baseline in total SOWS score will be presented for the Safety Analysis Set.

A figure for the SOWS scores over time will be created for all subjects in the Safety Analysis Set. An additional table and figure will be created for the Safety Analysis Set excluding subjects using illicit opioids (either by UDS or TLFB) at any time during the study.

## 9.5.4 Opioid Craving VAS Total Score

Opioid Craving VAS total scores will be summarized using descriptive statistics (mean, median, SD, minimum, and maximum), including change from baseline for the Safety Analysis Set. Additionally, separate listings for the actual values and the change from baseline in opioid craving VAS total scores will be presented for the Safety Analysis Set.



A figure for the Opioid Craving VAS scores over time will be created for all subjects in the Safety Analysis Set. An additional table and figure will be created for the Safety Analysis Set excluding subjects using illicit opioids (either by UDS or TLFB) at any time during the study.

## 9.6 Primary Safety Analyses

#### 9.6.1 Incidence of Adverse Events

#### 9.6.1.1 Adverse Events

#### Imputation of AE (for determination of TEAE only) and concomitant medication start and stop dates:

Start Date: If only 'day' is missing, and the month and year are not the same as the month of first dose, then impute day with '01'. Otherwise, if the month and year are the same as the first dose date, use the first dose date. If 'day' and 'month' are missing, and 'year' is not missing, then impute month and day with month and day of the first dose date (assuming same 'year'). If 'day' and 'month' are missing and 'year' is not missing and is not the same year as first dose date, then impute with '01' for both 'day' and 'month'. If the start date is completely missing, it will be set to the first dose date.

Stop Date: If only 'day' is missing, impute day with last day of the month. If 'day' and 'month' are missing, and 'year' is not missing, then impute month with '12' and day with '31' (or date of study discontinuation/completion if earlier than 12-31 and year is the same as the year of discontinuation). If the stop date is completely missing, it will be set to the date of study discontinuation/completion. A stop date will not be applied to ongoing AEs or ongoing medications.

#### **Treatment-related Adverse Events**

Any AE with a relationship to study treatment of 'Related' or missing will be considered a treatment-related AE as determined by the Investigator.

A summary of treatment-emergent AEs will be presented for the Safety Analysis Set and the Run-In Safety Analysis Set, including the number of events reported, the number and percentage of subjects reporting at least one AE, the number and percentage of subjects with the following:

- Related AEs
- SAEs
- Related SAEs
- AEs with an outcome of death
- Severe TEAEs
- AEs leading to discontinuation

A breakdown of the number and percentage of subjects reporting each AE categorized by SOC and PT coded according to the MedDRA dictionary version 17.1 will be presented for the Run-In period using the Run-In Safety Analysis Set and for the open label RBP-6000 treatment period using the Safety Analysis Set. Note that counting will be by subject not event and subjects are only counted once within each SOC or PT. AEs/TEAEs related to SUBOXONE/study treatment will presented in a similar manner.

A further tabulation of events experienced by ≥5% of subjects by SOC and PT will be presented for the Safety Analysis Set.

A summary of events reported, categorized by severity, will also be provided. Subjects with multiple events within a particular SOC or PT will be counted under the category of their most severe event within that SOC or PT. A further tabulation of severe AE/TEAEs will be presented by SOC and PT.

Additionally, treatment-related AEs/TEAEs will be summarized by maximum severity (Mild, Moderate, or Severe). A breakdown of severe treatment-related AEs/TEAEs by SOC and PT will be provided.

All AEs (including non-TEAEs) recorded on the CRF will be listed.

Statistical Analysis Plan

Effective Date: 10-Apr-2017 Version 3.0

Sponsor: Indivior Inc.
Protocol no: RB-US-13-0003

#### 9.6.1.2 Serious Adverse Events

SAEs and treatment-related SAEs will be summarized separately by SOC and PT for the Run-In Safety Analysis Set and the Safety Analysis Set.

All SAEs recorded on the CRF will be listed for all screened subjects.

#### 9.6.1.3 Adverse Events Leading to Discontinuation

A summary of AEs/TEAEs and treatment-related AEs/TEAEs leading to discontinuation (defined as an event with an outcome of 'drug withdrawn' in the CRF) will be provided, grouped by SOC and PT, for the Run-In Safety Analysis Set and the Safety Analysis Set. Supportive listings will be provided.

All AEs leading to discontinuation recorded on the CRF will be listed for the Run-In Safety Analysis Set and the Safety Analysis Set. Additionally, TEAEs leading to dose reduction will be listed for the Safety Analysis Set.

Additionally, TEAEs leading to dose reduction will be listed for the Safety Analysis Set

#### 9.6.1.4 Deaths

A table presenting the number and percentage of subjects who died during the Run-In period and during the open–label treatment period will be presented for the Run-In Safety Analysis Set, respectively. Deaths occurring in the study will also be listedfor all screened subjects.

#### 9.6.1.5 Potentially Pertaining to Drug Withdrawal Symptoms

A summary of TEAEs potentially pertaining to drug withdrawal, as defined in Appendix 2, will be summarized by SOC and PT for the Safety Analysis Set.

#### 9.6.1.6 Potentially Pertaining to Pancreatitis

A summary of TEAEs potentially pertaining to pancreatitis, as defined in <u>Appendix 2</u>, will be summarized by SOC and PT for the Safety Analysis Set.

#### 9.6.1.7 Potentially Pertaining to Hepatic Disorders

A summary of TEAEs potentially pertaining to hepatic disorders, as defined in <a href="Appendix 2">Appendix 2</a>, will be summarized by SOC and PT for the Safety Analysis Set.

#### 9.6.1.8 Potentially Pertaining to Injection Site Reactions

A summary of TEAEs potentially pertaining to injection site reactions, as defined in <u>Appendix 2</u>, will be summarized by SOC and PT for the Safety Analysis Set.

#### 9.6.1.9 Potentially Pertaining to Respiratory Depression and Failure

A summary of TEAEs potentially pertaining to respiratory depression and failure, as defined in Appendix 2, will be summarized by SOC and PT for the Safety Analysis Set.

#### 9.6.1.10 Potentially Pertaining to Central Nervous System Depression

A summary of TEAEs potentially pertaining to central nervous system depression, as defined in <u>Appendix 2</u>, will be summarized by SOC and PT for the Safety Analysis Set.

#### 9.6.1.11 Potentially Pertaining to Orthostatic Hypotension

A summary of TEAEs potentially pertaining to orthostatic hypotension, as defined in <u>Appendix 2</u>, will be summarized by SOC and PT for the Safety Analysis Set.



#### 9.6.2 Laboratory Data

Laboratory data will be reported using International System (SI) units as collected by the central laboratory. Unless otherwise specified, all continuous laboratory data will be summarized using descriptive statistics (n, mean, SD, median, min, and max) for each scheduled study assessment as well as change from baseline and percentage change from baseline [if applicable] by parameter class (hematology, chemistry, and urinalysis). The following parameters will have graphs of the mean values by visit through the end of study: hematocrit, alkaline phosphatase (ALP), alanine aminotransferase (ALT), amylase, lipase, trypsinogen, aspartate aminotransferase (AST), creatinine clearance, creatinine kinase, gamma-glutamyl transferase, and bilirubin (from serum chemistry results). All laboratory assessments include a baseline summary as defined in <a href="Section 5">Section 5</a> unless otherwise indicated. Hematology, chemistry, and urinalysis data will be summarized by displaying shifts from baseline value (low/normal/high) to last assessment on treatment and worst result on treatment (for only subjects with normal as baseline) considering both scheduled and unscheduled assessments. All laboratory assessments will be listed by panel with the corresponding normal ranges for each parameter. Screening laboratory will be provided in a separate listing.

#### 9.6.2.1 Hematology

Parameters include hematocrit, hemoglobin, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, mean corpuscular volume, platelet count, pancreatic enzymes, absolute red blood cell count, and absolute white blood cell count. Visits include Week 1 Day 1, Week 3 Day 15, Week 5 Day 29, Week 7 Day 43, Week 9 Day 57, Week 11 Day 71, Week 13 Day 85, Week 15 Day 99, Week 17 Day 113, Week 19 Day 127, Week 21 Day 141, Week 25 Day 169, Week 29 Day 197, Week 33 Day 225, Week 37 Day 253, Week 41 Day 281, Week 45 Day 309, Week 49 Day 337, and end of study visit.

#### 9.6.2.2 Serum Chemistry

Parameters include albumin, ALP, ALT, amylase, AST, blood urea nitrogen, calcium, calculated creatinine clearance, carbon dioxide, chloride, creatinine, creatinine kinase and subtypes, gamma-glutamyl transferase, globulin, glucose (non-fasting), high-density lipoprotein, immunoreactive trypsinogen, lactate dehydrogenase, lipase, low-density lipoprotein, magnesium, phosphorus, potassium, sodium, total bilirubin, direct bilirubin, total cholesterol, total protein, triglycerides, and uric acid. Visits include Week 1 Day 1, Week 3 Day 15, Week 5 Day 29, Week 7 Day 43, Week 9 Day 57, Week 11 Day 71, Week 13 Day 85, Week 15 Day 99, Week 17 Day 113, Week 19 Day 127, Week 21 Day 141, Week 25 Day 169, Week 29 Day 197, Week 33 Day 225, Week 37 Day 253, Week 41 Day 281, Week 45 Day 309, Week 49 Day 337, and end of study visit.

An additional summary of potential hepatotoxicity will be presented with the number and percentage of subjects at each time point and at any point on study that meet the following conditions: ALT > 3 × upper limit of normal (ULN), ALT >= 3 × ULN to <5 × ULN, ALT >= 5 × ULN to <8 × ULN, ALT >= 8 × ULN, AST > 3 × ULN, AST >= 3 × ULN to <5 × ULN, AST >= 5 × ULN to <8 × ULN, AST >= 8 × ULN, ALT > 3 × ULN and AST >= 3 × ULN, ALT and AST >= 3 × ULN to <5 × ULN, ALT and AST >= 5 × ULN to <5 × ULN, Bilirubin >= 5 × ULN to <5 × ULN, Bilirubin >= 5 × ULN Hy's Law cases which is defined as AST > 3 × ULN or ALT > 3 × ULN, bilirubin > 2 × ULN, and ALP <2 × ULN, and Modified Hy's Law which is defined as AST > 3 × ULN **AND** ALT > 3 × ULN, bilirubin > 2 × ULN, and ALP <2 × ULN. A listing of these cases including the results for the parameters and the number of times the ULN each result is will be provided. Figures of ALT [× ULN] vs. total bilirubin [× ULN] and AST [× ULN] vs. total bilirubin [× ULN] on a log/log scale and box plots of AST, ALT, and total bilirubin will be presented

An additional summary of high values of amylase, lipase, and trypsinogen will be presented with the number and percentage of subjects at each time point and at any point on study that meet the following conditions: Amylase > 3 × upper limit of normal (ULN), Lipase > 3 × ULN, and Trypsinogen> ULN. A listing of these cases including the results for the parameters and the number of times the ULN each result is will be provided.



#### 9.6.2.3 Urinalysis

Parameters include appearance, bilirubin, color, glucose, ketones, leucocyte esterase, nitrite, occult blood, pH, protein, specific gravity, and urobilinogen.

#### 9.6.2.4 Urine Drug Screen

Parameters include: opioids, cocaine, amphetamines, methadone, cannabinoids, barbiturates, benzodiazepines, methamphetamine, and phencyclidine. All drugs detected in the urine drug screen will be listed.

#### 9.6.3 Vital Signs

Measurements of vital signs (blood pressure systolic, blood pressure diastolic, pulse rate, oral temperature, pulse oximetry, weight, height, BMI, and waist-to-hip ratio) will be summarized using descriptive statistics at each scheduled visit and time point including change from baseline and percentage change from baseline.

Listings of all vital sign assessments will be provided in the following groups:

- Blood pressure systolic, blood pressure diastolic, pulse rate, oral temperature, and respiration rate
- Pulse Oximetry
- Body weight, BMI, and waist-to-hip ratio.

#### 9.6.4 Other Safety Variables

#### 9.6.4.1 12-lead Electrocardiograms

Results from 12-lead ECGs as determined by central reader will be categorized as normal or abnormal and will be summarized using shift from baseline to end of study/early termination using frequency counts. An additional table summarizing shift from baseline to worst result on study will be presented. ECG interval measurements including change from baseline will be summarized by time point using descriptive statistics for actual value and change from baseline. Parameters will include heart rate (beats/min), PR Interval (msec), QRS Duration (msec), RR interval (msec), QT interval (msec), adjudicated QTc-Bazett (msec), and adjudicated QTc-Fridericia (msec). Additionally, the number and percentage of subjects with a >30 msec or >60 msec change from baseline will be summarized by visit and at any point throughout the study. ECG results will be listed for interpretation and for the interval measurements.

#### 9.6.4.2 Suicidality

Suicidal ideation and suicidal behavior responses (Yes/No) will be summarized using counts and percentages in the Safety Analysis Set. Shift tables to demonstrate changes in eC-SSRS categories and changes in suicidal ideation and behavior scores, as defined in Section 5 from baseline during the openlabel treatment period will be presented. eC-SSRS and suicidal ideation responses will be listed separately. The suicidal ideation intensity ratings, each of the five items and the total score of the intensity for subjects with an ideation will be listed.

Several subjects completed the baseline-lifetime version of the e-CSSRS questionnaire that was intended to be used at Screening rather than the 'since last visit' version required at all subsequent visits. The data collected using the wrong version will be presented in the listings, but will not presented in the summary tables.

#### 9.6.4.3 Local Injection Site Tolerability

Local injection site tolerability as assessed by the Injection Site Grading scale will be summarized by category (pain, tenderness, erythema/redness, induration, and swelling) and severity at each time point and at any time using frequency counts and percentages.

Statistical Analysis Plan

Effective Date: 10-Apr-2017 Version 3.0

Sponsor: Indivior Inc.
Protocol no: RB-US-13-0003

A separate listing will be presented for severe/life threatening responses with their corresponding VAS scores.

The injection site tolerability results will be listed.

#### 9.6.4.4 Injection Site Pain

Injection Site Pain VAS scores will be summarized by subject type, injection, and time point after injection. The burning/stinging categorical variable (Yes/No) will be summarized by percentage of responses in each subject type at each time point. Attempted removal results will be summarized by percentage of subjects with attempted removal in each subject type at each visit.

Separate listings for burning/stinging and attempted removal evaluations will be provided. A listing of injection site pain VAS scores will also be provided.

#### 9.6.4.5 Other Safety Variables

Urine pregnancy results will be listed.

## 9.7 Pharmacokinetic Analysis

A listing of the PK data, including buprenorphine and norbuprenorphine plasma concentration measurement, will be provided. The population PK analysis of the drug plasma concentration data will be reported separately.

#### 10.0 Validation

PRA's goal is to ensure that each TFL delivery is submitted to the highest level of quality. Our quality control procedures will be documented separately in the study specific quality control plan.

#### 11.0 References

United States Department of Health and Human Services: Food and Drug Administration. Guidance for Industry: E14 Clinical Evaluation of QT/QTc Interval Prolongation and Proarrhythmic Potential for Non-Antiarrhythmic Drugs. October 2005.

PRS 005 T 17 E 



## **Appendix 1 Glossary of Abbreviations**

| Glossary of Abbreviations: | |
|---|---|
| ADY Analysis Day | |
| AE | Adverse event |
| ALP | Alkaline Phosphatase |
| ALT | Alanine Aminotransferase |
| AST | Aspartate Aminotransferase |
| BMI | Body Mass Index |
| CDF | Cumulative Distribution Function |
| CRF | Case Report Form |
| cows | Clinical Opioid Withdrawal Scale |
| CTMS | Clinical Trials Management System |
| eC-SSRS | Electronic Columbia Suicide Severity Rating Scale |
| | Electrocardiogram |
| ECG | End of Study |
| | · |
| ET | Early Termination Interim Analysis |
| IA | - |
| IDC<br>MadDDA | Individual Drug Counseling Medical Distinguishers Activities |
| MedDRA | Medical Dictionary for Regulatory Activities Protocol Deviation |
| PDV | |
| PK | Pharmacokinetic |
| PT | Preferred Term |
| RBP | Reckitt Benckiser Pharmaceuticals Inc. |
| SAP | Statistical Analysis Plan |
| SAE | Serious Adverse Event |
| SC | Subcutaneous |
| SD | Standard Deviation |
| SDTM | Study Data Tabulation Model |
| SDTMIG | Study Data Tabulation Model Implementation Guide |
| SI | International System |
| SOC | System Organ Class |
| SOWS | Subjective Opioid Withdrawal Scale |
| TEAE | Treatment-Emergent Adverse Event |
| TLFB | Timeline Followback |



| TFLs | Tables, Listings, and Figures |
|---------|-------------------------------------------|
| UDS | Urine Drug Screen |
| ULN | Upper Limit of Normal |
| VAS | Visual Analog Scale |
| WHODRUG | World Health Organization Drug Dictionary |



# Appendix 2 List of Preferred Terms from Standard MedDRA Queries for Adverse Events of Special Interest

## **Adverse Events Potentially Pertaining to Pancreatitis**

| Preferred Terms Potentially Pertaining to Pancreatitis | | |
|---|---|---|
| Amylase abnormal | Hyperbilirubinaemia | Pancreatic haemorrhage |
| Amylase creatinine clearance ratio abnormal | Hyperlipasaemia | Pancreatic necrosis |
| Amylase increased | Ischaemic pancreatitis | Pancreatic phlegmon |
| Bilirubin conjugated abnormal | Lipase abnormal | Pancreatic pseudocyst |
| Blood bilirubin increased | Lipase increased | Pancreatic pseudocyst drainage |
| Blood trypsin increased | Lipase urine increased | Pancreatitis |
| Cullen's sign | Oedematous pancreatitis | Pancreatitis acute |
| Grey Turner's sign | Pancreatic abscess | Pancreatitis haemorrhagic |
| Haemorrhagic necrotic pancreatitis | Pancreatic enzyme abnormality | Pancreatitis necrotising |
| Hereditary pancreatitis | Pancreatic enzymes abnormal | Pancreatitis relapsing |
| Hyperamylasaemia | Pancreatic enzymes increased | Pancreatorenal syndrome |

#### Adverse Events Potentially Pertaining to Respiration Depression and Failure

| Preferred Terms Potentially Pertaining to Respiratory Depression and Failure | | |
|---|---|---|
| Acute respiratory distress syndrome | Hypopnoea | Respiratory depression |
| Acute respiratory failure | Hypoventilation | Respiratory depth decreased |
| Apnoea | Hypoventilation neonatal | Respiratory distress |
| Apnoea neonatal | Lung hypoinflation | Respiratory failure |
| Infantile apnoea | Meconium aspiration syndrome | Respiratory paralysis |
| Apnoeic attack | Neonatal respiratory arrest | Respiratory rate decreased |
| Bradypnoea | Neonatal respiratory depression | Severe acute respiratory syndrome |
| Breath sounds absent | Neonatal respiratory distress syndrome | Cardio-respiratory arrest |
| Cardio-respiratory distress | Neonatal respiratory failure | Cardio-respiratory arrest neonatal |
| Central-alveolar hypoventilation | Respiratory arrest | Cardiopulmonary failure |
| Chronic respiratory failure | | |



## Adverse Events Potentially Pertaining to Central Nervous System Depression

| Preferred Terms Potenti | ally Pertaining to Central Nervous | System Depression |
|---|---|---|
| Mental fatigue | Postictal state | Psychomotor seizures |
| Microsleep | Consciousness fluctuating | Simple partial seizures |
| Narcolepsy | Neonatal oversedation | Autonomic seizure |
| Coma | Hypoglycaemic unconsciousness | Atonic seizures |
| Impaired driving ability | Hyperglycaemic unconsciousness | Seizure |
| Impaired ability to use machinery | Post-injection delirium sedation syndrome | Partial seizures with secondary generalisation |
| Accident | Preictal state | Alcoholic seizure |
| Road traffic accident | Psychogenic pseudosyncope | Partial seizures |
| Vision blurred | Mental status changes | Seizure like phenomena |
| Vertigo CNS origin | Mental status changes postoperative | Seizure cluster |
| Incoherent | Slow response to stimuli | Change in seizure presentation |
| Disturbance in attention | Unresponsive to stimuli | Migraine-triggered seizure |
| Judgement impaired | Hyporesponsive to stimuli | Psychogenic seizure |
| Mental impairment | Benign familial neonatal convulsions | Seizure anoxic |
| Borderline mental impairment | Febrile convulsion | Post stroke seizure |
| Cognitive disorder | Drug withdrawal convulsions | Accidental death |
| Altered state of consciousness | Convulsion neonatal | Accidental overdose |
| Depressed level of consciousness | Convulsions local | Accidental exposure to product |
| Lethargy | Tonic convulsion | Cerebrovascular accident |
| Loss of consciousness | Convulsion in childhood | Dizziness |
| Sedation | Clonic convulsion | Dizziness exertional |
| Somnolence | Acute encephalitis with refractory, repetitive partial seizures | Dizziness postural |
| Somnolence neonatal | Generalised tonic-clonic seizure | Procedural dizziness |
| Stupor | Complex partial seizures | Neurotoxicity |
| Syncope | | |

## **Adverse Events Potentially Pertaining to Orthostatic Hypotension**

| Preferred Terms Potentially Pertaining to Orthostatic Hypotension | | |
|---|---|---|
| Orthostatic hypotension | Vision blurred | Dizziness |
| Dizziness exertional | Dizziness postural | Syncope |
| Presyncope | Diastolic hypotension | Hypotension |

PRS 005 T 17 E 



## **Adverse Events Potentially Pertaining to Drug Withdrawal Symptoms**

| Preferred Terms Potentially Pertaining to Drug Withdrawal Symptoms | | |
|---|---|---|
| Agitation | Hypertension | Piloerection |
| Anxiety | Hypervigilance | Pruritus |
| Arthralgia | Influenza like illness | Psychomotor hyperactivity |
| Bone pain | Insomnia | Pyrexia |
| Chills | Irritability | Respiratory rate increased |
| Decreased appetite | Lacrimal disorder | Restlessness |
| Depression | Lacrimation increased | Rhinitis |
| Diarrhoea | Malaise | Rhinorrhoea |
| Dizziness | Muscle spasms | Sneezing |
| Drug dependence | Muscle twitching | Tachycardia |
| Flushing | Myalgia | Tremor |
| Heart rate increased | Mydriasis | Vomiting |
| Hyperhidrosis | Nausea | Yawning |
| Drug Withdrawal Syndrome | | |

## **Adverse Events Potentially Pertaining to Hepatic Events**

| Preferred Terms Potentially Pertaining to Hepatic Events | | |
|---|---|---|
| Bilirubin excretion disorder | Oesophageal varices | Galactose elimination capacity |
| | haemorrhage | test decreased |
| Cholaemia | Peripancreatic varices | Gamma-glutamyltransferase |
| | | abnormal |
| Cholestasis | Portal fibrosis | Gamma-glutamyltransferase |
| | | increased |
| Cholestatic liver injury | Portal hypertension | Guanase increased |
| Cholestatic pruritus | Portal hypertensive enteropathy | Hepaplastin abnormal |
| Drug-induced liver injury | Portal hypertensive gastropathy | Hepaplastin decreased |
| Hepatitis cholestatic | Portal vein cavernous | Hepatic artery flow decreased |
| | transformation | |
| Hyperbilirubinaemia | Portal vein dilatation | Hepatic congestion |
| Icterus index increased | Portopulmonary hypertension | Hepatic enzyme abnormal |
| Jaundice | Renal and liver transplant | Hepatic enzyme decreased |
| Jaundice cholestatic | Retrograde portal vein flow | Hepatic enzyme increased |
| Jaundice hepatocellular | Reye's syndrome | Hepatic function abnormal |
| Mixed liver injury | Reynold's syndrome | Hepatic hydrothorax |
| Ocular icterus | Splenic varices | Hepatic hypertrophy |
| Parenteral nutrition associated | Splenic varices haemorrhage | Hepatic mass |
| liver disease | | |
| Deficiency of bile secretion | Steatohepatitis | Hepatic pain |
| Yellow skin | Subacute hepatic failure | Hepatic sequestration |
| Acute hepatic failure | Varices oesophageal | Hepatic vascular resistance |
| | | increased |





| Acute on chronic liver failure | Varicose veins of abdominal wall | Hepatobiliary scan abnormal |
|---|---|---|
| Acute yellow liver atrophy | Anorectal varices | Hepatomegaly |
| Ascites | Anorectal varices haemorrhage | Hepatosplenomegaly |
| Asterixis | Intrahepatic portal hepatic venous fistula | Hyperammonaemia |
| Bacterascites | Peritoneovenous shunt | Hyperbilirubinaemia |
| Biliary cirrhosis | Portal shunt | Hypercholia |
| Biliary cirrhosis primary | Portal shunt procedure | Hypertransaminasaemia |
| Biliary fibrosis | Small-for-size liver syndrome | Kayser-Fleischer ring |
| Cholestatic liver injury | Spider naevus | Liver function test abnormal |
| Chronic hepatic failure | Splenorenal shunt | Liver induration |
| Coma hepatic | Splenorenal shunt procedure | Liver palpable |
| Cryptogenic cirrhosis | Spontaneous intrahepatic portosystemic venous shunt | Liver scan abnormal |
| Diabetic hepatopathy | Stomal varices | Liver tenderness |
| Drug-induced liver injury | Acute graft versus host disease in | Mitochondrial aspartate |
| - | liver | aminotransferase increased |
| Duodenal varices | Allergic hepatitis | Molar ratio of total branched- |
| | | chain amino acid to tyrosine |
| Gallbladder varices | Autoimmune hepatitis | Oedema due to hepatic disease |
| Gastric variceal injection | Chronic graft versus host disease in liver | Perihepatic discomfort |
| Gastric variceal ligation | Chronic hepatitis | Retrograde portal vein flow |
| Gastric varices | Graft versus host disease in liver | Total bile acids increased |
| Gastric varices haemorrhage | Hepatitis | Transaminases abnormal |
| Hepatectomy | Hepatitis acute | Transaminases increased |
| Hepatic atrophy | Hepatitis cholestatic | Ultrasound liver abnormal |
| Hepatic calcification | Hepatitis chronic active | Urine bilirubin increased |
| Hepatic cirrhosis | Hepatitis chronic persistent | X-ray hepatobiliary abnormal |
| Hepatic encephalopathy | Hepatitis fulminant | 5'nucleotidase increased |
| Hepatic encephalopathy | Hepatitis toxic | Blood alkaline phosphatase |
| prophylaxis | | abnormal |
| Hepatic failure | Ischaemic hepatitis | Blood alkaline phosphatase increased |
| Hepatic fibrosis | Lupus hepatitis | Blood cholinesterase abnormal |
| Hepatic hydrothorax | Non-alcoholic steatohepatitis | Blood cholinesterase decreased |
| Hepatic infiltration eosinophilic | Radiation hepatitis | Deficiency of bile secretion |
| Hepatic lesion | Steatohepatitis | Glutamate dehydrogenase increased |
| Hepatic necrosis | Granulomatous liver disease | Haemorrhagic ascites |
| Hepatic steato-fibrosis | Liver sarcoidosis | Hepatic fibrosis marker abnormal |
| Hepatic steatosis | Portal tract inflammation | Hepatic fibrosis marker increased |
| Hepatitis fulminant | Alanine aminotransferase abnormal | Hypoalbuminaemia |
| Hepatobiliary disease | Alanine aminotransferase increased | Leucine aminopeptidase increased |
| Hepatocellular foamy cell syndrome | Ammonia abnormal | Liver function test decreased |
| Hepatocellular injury | Ammonia increased | Liver function test increased |





| Hepatopulmonary syndrome | Ascites | Liver iron concentration |
|---|---|---|
| 16.7 | | abnormal |
| Hepatorenal failure | Aspartate aminotransferase | Liver iron concentration |
| | abnormal | increased |
| Hepatorenal syndrome | Aspartate aminotransferase | Model for end stage liver |
| | increased | disease score abnormal |
| Hepatotoxicity | Bacterascites | Model for end stage liver |
| | | disease score increased |
| Intestinal varices | Bile output abnormal | Periportal oedema |
| Intestinal varices haemorrhage | Bile output decreased | Peritoneal fluid protein abnormal |
| Liver and small intestine | Biliary ascites | Peritoneal fluid protein |
| transplant | | decreased |
| Liver dialysis | Bilirubin conjugated abnormal | Peritoneal fluid protein increased |
| Liver disorder | Bilirubin conjugated increased | Pneumobilia |
| Liver injury | Bilirubin urine present | Portal vein flow decreased |
| Liver operation | Biopsy liver abnormal | Portal vein pressure increased |
| Liver transplant | Blood bilirubin abnormal | Retinol binding protein |
| | | decreased |
| Lupoid hepatic cirrhosis | Blood bilirubin increased | Urobilinogen urine decreased |
| Minimal hepatic encephalopathy | Blood bilirubin unconjugated increased | Urobilinogen urine increased |
| Mixed liver injury | Bromosulphthalein test abnormal | Alcoholic liver disease |
| Nodular regenerative | Child-Pugh-Turcotte score | Cirrhosis alcoholic |
| hyperplasia | abnormal | |
| Non-alcoholic fatty liver | Child-Pugh-Turcotte score | Fatty liver alcoholic |
| ĺ | increased | ' |
| Non-alcoholic steatohepatitis | Computerised tomogram liver | Hepatic steato-fibrosis |
| Non-cirrhotic portal | Foetor hepaticus | Hepatitis alcoholic |
| hypertension | | |
| Oedema due to hepatic disease | Galactose elimination capacity | Zieve syndrome |
| | test abnormal | |



## Adverse Events Potentially Pertaining to Injection Site Reactions

| Preferred Terms Potentially Pertaining to Injection Site Reactions | | |
|---|---|---|
| Immediate post-injection | Injection site irritation | Injection site movement |
| reaction | | impairment |
| Injection related reaction | Injection site mass | Injection site lymphadenopathy |
| Injection site abscess | Injection site necrosis | Injection site nodule |
| Injection site cellulitis | Injection site nerve damage | Embolia cutis medicamentosa |
| Injection site infection | Injection site oedema | Injection site scar |
| Injection site pustule | Injection site pain | Injection site discharge |
| Injection site abscess sterile | Injection site paraesthesia | Injection site pallor |
| Injection site anaesthesia | Injection site phlebitis | Injection site papule |
| Injection site atrophy | Injection site pruritus | Injection site injury |
| Injection site bruising | Injection site rash | Injection site scab |
| Injection site cyst | Injection site reaction | Injection site eczema |
| Injection site dermatitis | Injection site thrombosis | Injection site streaking |
| Injection site erosion | Injection site ulcer | Injection site dryness |
| Injection site erythema | Injection site urticaria | Injection site laceration |
| Injection site extravasation | Injection site vesicles | Injection site macule |
| Injection site fibrosis | Injection site warmth | Injection site vasculitis |
| Injection site granuloma | Injection site ischaemia | Injection site exfoliation |
| Injection site haematoma | Injection site coldness | Injection site dysaesthesia |
| Injection site haemorrhage | Injection site discolouration | Injection site plaque |
| Injection site hypersensitivity | Injection site photosensitivity | Injection site hyperaesthesia |
| | reaction | |
| Injection site hypertrophy | Injection site swelling | Injection site hypoaesthesia |
| Injection site induration | Injection site discomfort | Injection site hypertrichosis |
| Injection site inflammation | Injection site calcification | |



# Appendix 3 List of Post-text Tables, Figures, Listings, and Supportive SAS Output Appendices

The TFL shells and table of contents for this study are provided in a separate document titled "Indivior 130003 SAP TFLs Version 3.0".